CLINICAL TRIAL: NCT00378963
Title: Instrument Applied and Manual Manipulation Induced EMG Response in Asymptomatic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: RD0606060022
Record Dates: First submitted 2006-09-18; First posted 2006-09-21 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-05

CONDITIONS: EMG Response

INTERVENTIONS:
Device: ProAdjuster

SUMMARY:
The purpose of this study is to determine the affects of instrumental and manual manipulation on the EMG response of asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic subjects (without somatosensory peripheral pain) will be recruited in the study. Subjects must sign an informed consent.

Exclusion Criteria:

Subjects with heart failure and any nervous system diseases will be excluded from the study. Additional exclusions include osteoporosis, diabetes, pregnancy, vascular insufficiency, and history of joint replacement therapy. Subjects under medical treatment, surgery and trauma within six months will be excluded.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Sung PS, Kang YM, Pickar JG. Effect of spinal manipulation duration on low threshold mechanoreceptors in lumbar paraspinal muscles: a preliminary report. Spine (Phila Pa 1976). 2005 Jan 1;30(1):115-22. doi: 10.1097/01.brs.0000147800.88242.48. PMID 15626991
- See also: Related Info — http://www.biopac.com